CLINICAL TRIAL: NCT02740660
Title: Effect on Body Composition With Albuterol and Caffeine Versus Placebo in Adolescents: A Pilot Study
Brief Title: Body Composition Changes With Albuterol and Caffeine Versus Placebo in Adolescents
Acronym: CAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Leverage Innovation for Technology Transfer Fund (LSU LIFT2) (Unknown)
Responsible Party: Principal Investigator, Daniel Hsia, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBRC 2015-065
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Pediatric Obesity
Keywords: Albuterol; Caffeine; Lean Body Mass; Fat Mass
MeSH Terms: conditions — Pediatric Obesity | interventions — Caffeine; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine 100mg / Albuterol 4mg (Experimental): One capsule 3 times per day orally for a total of 8 weeks and family weight management counseling for a total of 8 weeks.
  Interventions: Drug: Caffeine 100mg / Albuterol 4mg; Behavioral: Family weight management counseling
- Placebo (Placebo Comparator): One capsule 3 times per day orally for a total of 8 weeks and family weight management counseling for a total of 8 weeks.
  Interventions: Drug: Placebo; Behavioral: Family weight management counseling

INTERVENTIONS:
Drug: Caffeine 100mg / Albuterol 4mg
  Arms: Caffeine 100mg / Albuterol 4mg
Drug: Placebo
  Arms: Placebo
Behavioral: Family weight management counseling

SUMMARY:
The purpose of this study is to determine whether taking a combination of caffeine and albuterol three times per day will increase muscle and decrease fat in your child's body and to determine how these medications make your child feel. Albuterol is approved by the FDA for the treatment of asthma. It is not approved to increase muscle and decrease body fat in children.

DETAILED DESCRIPTION:
Previous studies done at Pennington Biomedical have demonstrated that the equivalent of oral albuterol 4mg three times a day (tid) with oral caffeine 100mg tid reduces body fat and increases lean tissue in rodents more than the addition of the effect of the two components separately. The combination of albuterol with caffeine changed body composition without changing food intake. An adult male taking albuterol 4 mg orally tid plus caffeine 100mg orally tid increased lean mass by 1.25% and decreased fat mass by 1.2% over a two month period. These effects are expected to be even greater in a growing adolescent. This pilot project will take the first step towards trying to understanding the safety and potential efficacy of this drug combination. The prospect of using inexpensive medications already approved in the pediatric population for the treatment of asthma as a novel treatment for adolescent obesity addresses a medical need that is presently unmet.

Food restriction in adolescence is not only difficult to accomplish, but it also raises concerns about growth and development. A medication approved for the treatment of obesity in the adolescent age group that improves body composition by reducing body fat and increasing lean tissue without needing to restrict food intake would be a useful tool for physicians who address the treatment of obesity in adolescents. Albuterol is a medication, approved for ages 6 and older, used for the treatment of asthma and has also been shown to increase muscle strength and lean body mass in children with spinal muscular atrophy and in healthy young men during an exercise training program. A drug approved for the treatment of adolescent obesity that increases lean tissue, decreases fat tissue and can be given in conjunction with lifestyle modifications would be welcomed by both pediatricians who treat these adolescents and by adolescents who are stigmatized by their obesity.

A provisional patent has been submitted by Pennington Biomedical Research Center to protect the combination of caffeine and albuterol in a 1:25 ratio for synergistically increasing muscle mass and decreasing fat mass as a potential treatment for obesity in adolescents.

This study will be a double-blinded, randomized, placebo-controlled, pilot study in which subjects will be randomized to receive either placebo or a combination of Albuterol 4 mg and Caffeine 100mg three times per day orally for a total of 8 weeks. Each subject will continue on the study intervention for the entire duration of treatment

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females with a BMI ≥ 95th percentile
* Between 12 and 17 years of age inclusive
* Tanner Stage III and above

Exclusion Criteria:

* Weigh less than 50 kg
* Have a family history of sudden death or hypertrophic cardiomyopathy
* Have a history of unexplained syncope
* Have a marked baseline prolongation of QT/QTc interval (QTc interval >450 ms), a history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or use concomitant medications that prolong the QT/QTc interval
* Have history of asthma, hypertension, thyroid disease, or significant neurologic disease such as seizure disorder
* Are pregnant, planning to become pregnant, or nursing. Females who are sexually active must be using adequate contraception.
* Take a medication known to affect weight or body composition like systemic glucocorticoids, atypical anti-psychotics, or weight loss medications
* Take beta-stimulators or beta-blockers on a regular basis
* Take stimulants for attention deficit disorder
* Take monoamine oxidase inhibitors, tricyclic antidepressants, or diuretics
* Take any chronic medication that has not had a stable dose for 1 month or longer
* Have type 1 or type 2 diabetes
* Have any significant cardiac disease (such as heart failure, arrhythmias, or valve disease), uncontrolled pulmonary disease, chronic liver disease, chronic kidney disease, or chronic infectious disease
* Have any significant psychiatric illness that is unstable or untreated such as bipolar disorder, severe depression, or severe anxiety
* Have a history of suicidal ideation
* Have an allergy or hypersensitivity to albuterol
* Are unwilling to discontinue caffeine-containing products while in the study
* Are deemed unfit to participate in the study based on evaluation by the medical investigator

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-04; Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hsia, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu AG, Arceneaux KP 3rd, Chu JT, Jacob G Jr, Schreiber AL, Tipton RC, Yu Y, Johnson WD, Greenway FL, Primeaux SD. The effect of caffeine and albuterol on body composition and metabolic rate. Obesity (Silver Spring). 2015 Sep;23(9):1830-5. doi: 10.1002/oby.21163. Epub 2015 Aug 4. PMID 26239482
- [Background] Skura CL, Fowler EG, Wetzel GT, Graves M, Spencer MJ. Albuterol increases lean body mass in ambulatory boys with Duchenne or Becker muscular dystrophy. Neurology. 2008 Jan 8;70(2):137-43. doi: 10.1212/01.WNL.0000287070.00149.a9. Epub 2007 Oct 17. PMID 17942817
- [Background] Caruso JF, Hamill JL, De Garmo N. Oral albuterol dosing during the latter stages of a resistance exercise program. J Strength Cond Res. 2005 Feb;19(1):102-7. doi: 10.1519/R-14793.1. PMID 15705021

RESULTS

PARTICIPANT FLOW:
Groups:
- Caffeine 100mg / Albuterol 4mg: One capsule 3 times per day orally for a total of 8 weeks and family weight management counseling for a total of 8 weeks.
  Caffeine 100mg / Albuterol 4mg
  Family weight management counseling
- Placebo: One capsule 3 times per day orally for a total of 8 weeks and family weight management counseling for a total of 8 weeks.
  Placebo
  Family weight management counseling
Period: Overall Study
Arm/Group | Caffeine 100mg / Albuterol 4mg | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine 100mg / Albuterol 4mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1.5) | 15 (1.9) | 14 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Mass With Caffeine/Albuterol
Description: DXA Scan of obese adolescents
Time Frame: Baseline, Week 8
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Caffeine 100mg / Albuterol 4mg | Placebo
Number analyzed (Participants) | 6 | 6
kg | 0.97 (1.11) | -0.21 (1.41)

2. Primary Outcome: Change in Lean Mass With Caffeine/Albuterol
Description: DXA Scan of obese adolescents
Time Frame: Baseline, Week 8
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Caffeine 100mg / Albuterol 4mg | Placebo
Number analyzed (Participants) | 6 | 6
kg | 1.34 (1.22) | 0.88 (1.16)

3. Primary Outcome: Change in Weight With Caffeine/Albuterol
Time Frame: Baseline, Week 8
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Caffeine 100mg / Albuterol 4mg | Placebo
Number analyzed (Participants) | 6 | 6
kg | 2.57 (1.92) | 1.05 (2.19)

4. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Week 2, Week 4, Week 6, Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine 100mg / Albuterol 4mg | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 5 | 2

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were collected at Week 2, 4, 6, 8
Arm/Group | Caffeine 100mg / Albuterol 4mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine 100mg / Albuterol 4mg (N=6) | Placebo (N=6)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Toothache (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a pilot study with a small number of participants. Diet and physical activity was not controlled in this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT02740660/Prot_SAP_000.pdf